CLINICAL TRIAL: NCT03309267
Title: Serratus Anterior Plane Block Versus Intercostal Block For Postoperative Analgesia Following Thoracotomy
Brief Title: Serratus Anterior Plane Block Versus Intercostal Block
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Gözen Öksüz, Assistant Professor, Kahramanmaras Sutcu Imam University
Other Study IDs: 2017/14-18
Record Dates: First submitted 2017-10-06; First posted 2017-10-13 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Pain, Postoperative
Keywords: pain, thoracotomy
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intercostal block: Anesthesia induction was performed to all patients .At the end of the operation some patients were performed with intercostal block by the chest surgeon. For 24 hours postoperatively, tramadol was administered with patient-controlled analgesia (PCA) All patients were extubated after the operation and transferred to ICU.
  Interventions: Procedure: Intercostal block
- Serratus anterior plane block: Anesthesia induction was performed to all patients. At the end of the operation some patients were performed SAPB under Ultrasound guidance by the same anesthetist.For 24 hours postoperatively, tramadol was administered with patient-controlled analgesia (PCA) All patients were extubated after the operation and transferred to ICU.
  Interventions: Procedure: Serratus anterior plane block

INTERVENTIONS:
Procedure: Intercostal block — Intercostal block +patient controlled analgesia
  Groups: Intercostal block
Procedure: Serratus anterior plane block — Serratus anterior plane block+patient controlled analgesia
  Groups: Serratus anterior plane block

SUMMARY:
Pain after thoracotomy is the most severe pain experienced by the patient. Good pain control after the operation provides comfortable respiration and reduces the development of chronic pain and complications.

we aimed to compare SAPB with IBregarding postoperative visual analog scale (VAS) scores and analgesic consumption in patients undergoing thoracotomy operation.

DETAILED DESCRIPTION:
Patients who underwent thoracotomy operation in our hospital between May 2016 and June 2017 were examined. A retrospective evaluation was made of the data that was retrieved from the records of a total of 49 patients aged 18-75 years, ASA I-III, who were applied with Intercostal (IB) or Serratus anterior plane(SAPB) for a thoracotomy operation. The patient information was retrieved from the patient records and anesthesia block forms. The data were examined in respect of age, sex, height, weight, ASA, operation type, operating time, the amount of postoperative analgesic consumption, VAS at 1.,2.,4.,6.,12.,24. hours and complications (atelectasis, nausea, vomiting, hypotension and bradycardia).

Statistical analysis was performed using the SPSS program for Mac, version 17.0 (SPSS,Chicago,IL). Descriptive statistics are presented as mean and SD, and as the number of cases (n) and the corresponding percentage (%) for nominal variables. T tests were performed for normally continuous variables. The Mann-Whitney U test was used for non-parametric variables. A value of p < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Thoracotomy operation
2. a.Serratus anaterior plane block b.Intercostal block

Exclusion Criteria:

1. missing data
2. written consent
3. rethoracotomy

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Thoracotomy Operation
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2017-11-03 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesic consumption | up to 24 hour
  Postoperative analgesic consumption

SECONDARY OUTCOMES:
Visuel analog scala (VAS) | up to 24 hour
  1.,2.,4.,6.,12.,24. hour

OTHER OUTCOMES:
Complications | Postoperative 1 week
  Postoperative Complications

CONTACTS AND LOCATIONS:
Overall Officials: Gözen Öksüz, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- KahramanmarasSIU, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Okmen K, Okmen BM. The efficacy of serratus anterior plane block in analgesia for thoracotomy: a retrospective study. J Anesth. 2017 Aug;31(4):579-585. doi: 10.1007/s00540-017-2364-9. Epub 2017 Apr 26. PMID 28447227